CLINICAL TRIAL: NCT02368912
Title: A Double Blind, Randomized, Placebo-controlled, Ascending Single and Multiple Oral Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ASP1707 in Healthy Young and Elderly Male Subjects and in Healthy Pre-menopausal Female Subjects Including an Open-label Comparison of Pharmacokinetics Under Fasted and Fed Conditions in Healthy Young Male Subjects
Brief Title: A Study to Assess the Safety, Tolerability and Effects of Single and Multiple Ascending Doses of ASP1707 in Healthy Male and Pre-menopausal Female Subjects, Including a Comparison of the Effects Under Fasted and Fed Conditions in Healthy Young Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1707-CL-0001; 2010-018292-21 (EudraCT Number)
Record Dates: First submitted 2014-11-14; First posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Pharmacokinetics of ASP1707; Pharmacodynamics of ASP1707
Keywords: Phase 1; ASP1707; Dose escalation; Food effect; Maximum tolerated dose (MTD); Healthy subjects; Single ascending dose; Multiple ascending dose
MeSH Terms: interventions — opigolix

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- 1. Single ascending dose (SAD), ASP1707 dose levels 1-7 (Experimental): healthy young male
  Interventions: Drug: ASP1707 single dose of dose levels 1 -7
- 2. Single ascending dose (SAD), placebo dose levels 1-7 (Experimental): healthy young male
  Interventions: Drug: Placebo single dose of dose levels 1-7
- 3. Food effect (FE), ASP1707 fasted (Experimental): Fasted healthy young male
  Interventions: Drug: ASP1707 single dose fasted
- 4. Food effect (FE), ASP1707 fed (Experimental): Fed healthy young male
  Interventions: Drug: ASP1707 single dose fed
- 5. Multiple ascending dose (MAD), ASP1707 dose levels 1-4 (Experimental): healthy elderly male
  Interventions: Drug: ASP1707 multiple dose of dose levels 1-4
- 6. Multiple ascending dose (MAD), Placebo, dose levels 1-4 (Experimental): healthy elderly male
  Interventions: Drug: Placebo multiple dose of dose levels 1-4
- 7. Multiple ascending dose (MAD), ASP1707, dose levels 1-2 (Experimental): healthy pre-menopausal female
  Interventions: Drug: ASP1707 multiple dose of dose levels 1-2
- 8. Multiple ascending dose (MAD), Placebo dose levels 1-2 (Experimental): healthy pre-menopausal female
  Interventions: Drug: Placebo multiple dose of dose levels 1-2
- 9. Parallel multiple dose, ASP1707 dose levels 1-3 (Experimental): healthy pre-menopausal female
  Interventions: Drug: ASP1707 parallel multiple dose of dose levels 1-3
- 10. Parallel multiple dose, Placebo (Experimental): healthy pre-menopausal female
  Interventions: Drug: Placebo parallel multiple dose

INTERVENTIONS:
Drug: ASP1707 single dose of dose levels 1 -7 — Oral, dose escalation
  Arms: 1. Single ascending dose (SAD), ASP1707 dose levels 1-7
Drug: Placebo single dose of dose levels 1-7 — Oral, dose escalation, healthy young male
  Arms: 2. Single ascending dose (SAD), placebo dose levels 1-7
Drug: ASP1707 single dose fasted — Oral, healthy young male
  Arms: 3. Food effect (FE), ASP1707 fasted
Drug: ASP1707 single dose fed — Oral, healthy young male
  Arms: 4. Food effect (FE), ASP1707 fed
Drug: ASP1707 multiple dose of dose levels 1-4 — Oral, multiple dose escalation, healthy elderly male
  Arms: 5. Multiple ascending dose (MAD), ASP1707 dose levels 1-4
Drug: Placebo multiple dose of dose levels 1-4 — Oral, multiple dose escalation, healthy elderly male
  Arms: 6. Multiple ascending dose (MAD), Placebo, dose levels 1-4
Drug: ASP1707 multiple dose of dose levels 1-2 — Oral, multiple dose escalation, healthy pre-menopausal female
  Arms: 7. Multiple ascending dose (MAD), ASP1707, dose levels 1-2
Drug: Placebo multiple dose of dose levels 1-2 — Oral, multiple dose escalation, healthy pre-menopausal female
  Arms: 8. Multiple ascending dose (MAD), Placebo dose levels 1-2
Drug: ASP1707 parallel multiple dose of dose levels 1-3 — Oral, multiple dose, healthy pre-menopausal female
  Arms: 9. Parallel multiple dose, ASP1707 dose levels 1-3
Drug: Placebo parallel multiple dose — Oral, dose escalation, healthy pre-menopausal female
  Arms: 10. Parallel multiple dose, Placebo

SUMMARY:
This study consists of four parts:

Part 1 is a randomized, double-blind, placebo-controlled, single ascending dose study in healthy young male subjects to evaluate the safety, tolerability pharmacokinetics (PK) and effect on certain hormones and if possible to determine the highest well-tolerated dose of ASP1707 in healthy young male subjects under fasted conditions.

Part 2 is an open label, randomized crossover, single dose study to determine the effect of food on the pharmacokinetics of ASP1707and effect on certain hormones in healthy young male subjects.

Part 3 is a randomized, double-blind, placebo-controlled, multiple ascending dose study to evaluate the safety, tolerability and pharmacokinetics (PK) of ASP1707 in healthy elderly men and healthy premenopausal females, and to determine the effect on certain hormones in males. Age and gender is also evaluated.

Part 4 is a randomized, double-blind, placebo-controlled, parallel, multiple dose study to evaluate the safety, tolerability and PK of ASP1707, and its effect on certain hormones in healthy pre-menopausal female subjects.

DETAILED DESCRIPTION:
Part 1 comprises 7 dose groups of 8 healthy young male subjects. ASP1707 or matching placebo ( 3 to 1 ratio) is given as a single dose under fasted conditions.

The first group receives the lowest dose while the last group receives the highest dose.

Part 2 (Food-Effect) The group consists of 12 healthy young male subjects who receive two separate doses of ASP1707 under fasted or fed conditions. Half of the subjects are dosed first under fasted condition and half of them had first an FDA high-fat breakfast. Subjects receive the alternate treatment on the second occasion. Dosing is separated by at least 7 days or 7 times t1/2 (terminal elimination half-life) as assessed from Part 1.

Part 3 Comprises 4 dose groups of 12 healthy elderly men each, and two groups of 12 healthy premenopausal women. The latter are dosed ASP1707 or placebo in parallel to the 4 male groups. Subjects are fasted or fed depending on observations from Part 2.

Dose levels are defined after evaluating interim safety, tolerability and PK and PD results from Part 1. A lower maximum dose is used in women than in men, based on preclinical data. Dose escalation in the men is independent from dose escalation in the women. Women and men receive once-daily dosing;

Part 4 includes 4 groups, 1 placebo and 3 for ASP1707, each with 9 pre-menopausal women. Subjects in each dose group receive a fixed daily dose. Subjects are domiciled for various intervals during each of 3 menstrual cycles. Dosing occurs for 21 Days during the subjects' second menstrual cycle of the study (Day 1 of Period 2); fasted or fed depending on observations from Part 2.

ELIGIBILITY:
Inclusion Criteria:

Parts 1 & 2:

* Healthy young male subject aged 18 to 45 years inclusive
* Body Mass Index more than or equal to 18.5 and less than 30.0 kg/m2.
* Male subjects must be non-fertile, or must practice an adequate contraceptive method to prevent pregnancies.

Part 3:

* Healthy elderly male subject aged 55 years or older, or healthy pre-menopausal female subject aged 18 to 45 inclusive.
* Body Mass Index more than or equal to 18.5 and less than 30.0 kg/m2.
* Male subject must be non-fertile, or must practice adequate contraceptive methods.
* Female subjects must be of non-child bearing potential, i.e. surgically sterilized or practice adequate (double barrier) non-hormonal contraceptive methods.

Part 4:

* Healthy pre-menopausal female subject aged 18 to 45 inclusive.
* Body Mass Index more than or equal to 18.5 and less than 30.0 kg/m2.
* Female subjects must be of non-child bearing potential, i.e. surgically sterilized or practice adequate contraceptive methods.
* Females having a regular menstruation cycle with a duration between 25 up to 30 days.

Exclusion Criteria:

Parts 1 & 2:

* Male subjects with out-of-range Testosterone levels in serum at screening.
* Subjects with any history of cancer.
* Any of the liver function tests (i.e. ALT and AST) above the upper limit of normal.
* A QTc interval of > 430 ms after repeated measurements.
* Regular use of any inducer of metabolism (e.g. barbiturates, rifampin) in the 3 months prior to admission to the Clinical Unit.
* Positive serology test for HBsAg, anti HAV (IgM), anti-HCV or anti-HIV 1+2.

Part 3:

* Pregnancy within 6 months before screening assessment or breast feeding 3 months before screening.
* Male subjects with out-of-range T levels in serum at screening.
* Positive serology test for HBsAg, anti HAV (IgM), anti-HCV or anti-HIV 1+2.

Part 4:

* Pregnancy within 6 months before screening assessment or breast feeding 3 months before screening.
* Use of any hormonal interfering contraceptives in the 3 months before admission (for 3 consecutive menstruation cycles) OR any evidence of unovulatory menstrual cycles.
* Positive serology test for HBsAg, anti HAV (IgM), anti-HCV or anti-HIV 1+2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2010-06; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Safety assessed by nature, frequency and severity of adverse events | Screening to End of Study Visit (ESV) (up to Day 19 and up to Day 39)
  Respectively Part 1 and Part 3
Safety assessed by physical examination | Screening to End of Study Visit (ESV) (up to Day 19 and up to Day 39)
  Respectively Part 1 and Part 3
Safety assessed by vital signs | Screening to End of Study Visit (ESV) (up to Day 19 and up to Day 39)
  Respectively Part 1 and Part 3. Vital signs include blood pressure and pulse.
Safety assessed by safety laboratory tests | Screening to End of Study Visit (ESV) (up to Day 19 and up to Day 39)
  Respectively Part 1 and Part 3, Biochemistry, hematology, and urinalysis
Safety assessed by 12 lead electrocardiogram (ECG) | Screening to End of Study Visit (ESV) (up to Day 19 and up to Day 39)
  Respectively Part 1 and Part 3
Safety assessed by continuous cardiac monitoring (Holter) | Days -1 and 21
  Part 3
Pharmacokinetics (PK) of ASP1707 measured by area under the plasma concentration - time curve (AUC) extrapolated to time = infinity (AUCinf) in plasma | Pre-dose (Day 1) to Day 5
  Part 2
PK of ASP1707 measured by area under the plasma concentration-time curve (AUC) to time from the time of dosing to the last measurable concentration (AUClast) in plasma | Pre-dose (Day 1) to Day 5
  Part 2
PK of ASP1707 measured by time to reach quantifiable concentrations (tlag) in plasma | Pre-dose (Day 1) to Day 5
  Part 2
PK of ASP1707 measured by time to attain maximum concentration (tmax) in plasma | Pre-dose (Day 1) to Day 5
  Part 2
PK of ASP1707 measured by Cmax in plasma | Pre-dose (Day 1) to Day 5
  Part 2
PK of ASP1707 measured by terminal elimination half-life (t1/2) in plasma | Pre-dose (Day 1) to Day 5
  Part 2
PK of ASP1707 measured by apparent volume of distribution (Vz/F) in plasma | Pre-dose (Day 1) to Day 5
  Part 2
PK of ASP1707 measured by apparent clearance (CL/F) in plasma | Pre-dose (Day 1) to Day 5
  Part 2
PK of ASP1707 measured by amount excreted unchanged into urine (Ae) from time of dosing until last measurable concentration (Aelast) in urine | Pre-dose (Day 1) to Day 5
  Part 2
PK of ASP1707 measured by Ae extrapolated to time = infinity (Aeinf) in urine | Pre-dose (Day 1) to Day 5
  Part 2
PK of ASP1707 measured by Ae in % up to the collection time of the last measurable concentration (Aelast%) in urine | Pre-dose (Day 1) to Day 5
  Part 2
PK of ASP1707 measured by Ae in % extrapolated to time infinity (Aeinf%) in urine | Pre-dose (Day 1) to Day 5
  Part 2
PK of ASP1707 measured by renal clearance (CLR) in urine | Pre-dose (Day 1) to Day 5
  Part 2
Pharmacodynamics (PD) of ASP1707 measured by Cmax in plasma | Day -1 to day 15 for period 1, Day 7 to Day 15 for periods 2 and 3
  Part 4, period 1, 2 and 3. Estradiol (E2), Follicle-stimulating hormone (FSH) and Luteinizing Hormone (LH) levels
PD of ASP1707 measured by tmax in plasma | Day -1 to day 15 for period 1, Day 7 to Day 15 for periods 2 and 3
  Part 4, period 1, 2 and 3. E2, FSH and LH levels
PD of ASP1707 measured by average concentration (Cavg, day 7-15) in plasma | Pre-dose to Day 26
  Part 4, period 1, 2 and 3. E2, FSH and LH levels
PD of ASP1707 measured by average concentration (Cavg, day 5-19) in plasma | Pre-dose to Day 26
  Part 4, period 3. E2, FSH and LH levels
PD of ASP1707 measured by average concentration (Cavg, day 23-26) in plasma | Pre-dose to Day 26
  Part 4, period 2. E2, FSH and LH levels
PD of ASP1707 - maximal duration within therapeutic range | Pre-dose to Day 26
  Part 4, period 2. E2 levels
PD of ASP1707 - total duration within therapeutic range (20-50 pg/mL) | Pre-dose to Day 26
  Part 4, period 2. E2 levels
PD of ASP1707 - Time of onset therapeutic range | Pre-dose to Day 26
  Part 4, period 2. E2 levels
PD of ASP1707 - Time of offset therapeutic range | Pre-dose to Day 26
  Part 4, period 2. E2 levels
PD of ASP1707 - Time of start menstruation after last dose of study drug | Pre-dose to Day 26
  Part 4, period 3

SECONDARY OUTCOMES:
PK profile of ASP1707 in plasma and urine for Part 1 | Pre-dose (Day 1) to Day 5
  AUCinf, AUClast, tlag, tmax, Cmax, t1/2, Vz/F, CL/F, Aelast, Aeinf, Aelast%, Aeinf%, CLR
Safety profile assessed by nature, frequency and severity of adverse events, physical examination, vital signs, safety laboratory tests and 12 lead ECG | Screening to End of Study Visit (ESV) (Up to 31 days and up to 62 days)
  Respectively Part 2 and Part 4
PD profile of ASP1707 for Part 1 and Part 2 | Pre-dose (Day 1) to Day 12-19
  Testosterone (T), LH and FSH levels: Cmin, tmin, maximal %Reduction and T only: Number and percentage of subjects with T castration level (= T < 0.5 ng/mL) after single dose, Time of onset of T < 0.5 ng/mL after single dose, Duration of T <0.5 ng/mL after single dose
PD profile of ASP1707 for Part 3 | Pre-dose (Day 1) to Day 39
  T, LH and FSH levels: Cmin, tmin, maximal %Reduction T only: Number and percentage of subjects with T < 0.5 ng/mL at any time post-first dose, Number and percentage of subjects with T < 0.5 ng/mL after last dose, Number of subjects reaching T<0.5 ng/mL for ≥14 days, Day of onset of T < 0.5 ng/mL after multiple doses of ASP1707 (T < 0.5 ng/mL for the first time), Time of onset of T < 0.5 ng/mL after first dose, Duration of T < 0.5 ng/mL after single dose and during multiple dosing, Total duration, Maximal duration:Time from last dose to return to baseline levels for T, LH and FSH, Duration of T < 0.5 ng/mL after last dose
PK profile of ASP1707 in plasma and urine for Part 3 | Pre-dose (Day 1) to Day 25
  AUCinf, AUClast, tlag, tmax, Cmax, t1/2, Vz/F, CL/F, Aelast, Aeinf, Aelast%, Aeinf%, CLR, Ctrough, AUC during the time interval between consecutive dosing (AUCtau), Accumulation Ratio (Rac), Peak Trough Ratio (PTR), Ae during the time interval between consecutive dosing (Aetau), Aetau as percentage of total dose (Aetau%), Ae during the time interval between consecutive dosing (AUCtau), (AUC0-24h), Ae0-24h, Ae0-24h%
PK profile of ASP1707 in plasma and urine for Part 4 | Pre-dose (Day 23) to Day 25
  AUCtau, tmax, Cmax, t1/2, Vz/F, CL/F, CLR, Ctrough, PTR, Aetau, Aetau%,

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- SGS Life Science Services, Aster, Paris, France